CLINICAL TRIAL: NCT01452425
Title: In Vivo Optical Spectroscopy Monitoring in a New Model of Muscular Compartment Syndrome.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Forget Patrice, MD, Université Catholique de Louvain
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: B40320107753
Record Dates: First submitted 2011-10-11; First posted 2011-10-14 (Estimated); Results first posted 2014-12-22 (Estimated); Last update posted 2014-12-22 (Estimated); Status verified 2014-12

CONDITIONS: Human Volunteers
Keywords: Human volunteers
MeSH Terms: interventions — Tourniquets

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tourniquet (Experimental): Inflation of a tourniquet
  Interventions: Device: Tourniquet; Device: INVOS assessment; Device: EMG assessment

INTERVENTIONS:
Device: Tourniquet — Inflation of a tourniquet (pressure equal to the mean arterial pressure) obtaining a model of slight venous congestion and arterial hypoperfusion
Device: INVOS assessment — Near Infraread spectroscopy, non invasive
Device: EMG assessment — Electromyography, non invasive

SUMMARY:
Muscular compartment syndrome (MCS) is consecutive to an increase in intramuscular compartment pressures, and is a rare but serious postoperative complication.

The INVOS (In Vivo Optical Spectroscopy) monitors tissular oxygenation continuously and non-invasively.

The objective is to develop a model mimicking the physiopathology of MCS to assess the interest of the INVOS in this case.

DETAILED DESCRIPTION:
After inflation of a tourniquet (pressure equal to the mean arterial pressure, we will obtain a model of slight venous congestion and arterial hypoperfusion. A comparison will be made between INVOS monitoring, sensory deficits, pain, electromyography and invasive pressure.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* >18yr
* Informed consent
* Male

Exclusion Criteria:

* Neuropathies
* Vascular pathology
* Actual pain
* Anti-platelet or anticoagulant therapy
* Ipsilateral history of fracture

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrice Forget, M.D., Principal Investigator — UCL
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tourniquet
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Tourniquet: No adverse event
Arm/Group | Tourniquet
Number analyzed (Participants) | 10
Age, Customized [Mean (Standard Deviation); unit: years]
  age | 33 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 10

OUTCOME MEASURES:

1. Primary Outcome: Comparison Between INVOS Monitoring and Electromyography
Description: A comparison will be made between the INVOS monitoring and non invasive (transcutaneous) EMG monitoring (AP Block), to determine the accuracy of the INVOS monitoring to predict AP block.
  Measures were:
  [mean (SD)] INVOS (in %) value at baseline and at the time of the block
Time Frame: 45 minutes
Measure: Mean (Standard Deviation); unit: % of StcO2
Arm/Group | Tourniquet
Number analyzed (Participants) | 10
% of StcO2
  INVOS (Baseline) | 73 (9)
  INVOS (At time of the block) | 46 (11)

2. Primary Outcome: Intracompartmental Pressure (ICP)
Description: [mean (SD)] ICP (in mmHg), value at baseline and at the time of the block
Time Frame: 45 minutes
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Tourniquet
Number analyzed (Participants) | 10
mmHg
  ICP (Baseline) | 17 (9)
  ICP (At time of the block) | 70 (6)

ADVERSE EVENTS:
Arm/Group | Tourniquet
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes